CLINICAL TRIAL: NCT01565473
Title: PET Study of Biochemistry and Metabolism of the CNS: Parkinson Disease
Brief Title: PET Study of Non-Motor Symptoms of Parkinson Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, M.D., Ph.D., University of Michigan
Other Study IDs: P01NS015655 (NIH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson Disease
Keywords: non-motor symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson disease patients
- Healthy normal controls

SUMMARY:
This research plan is focused on neurochemical positron emission tomography (PET) studies of Parkinson disease (PD). PD is the most common neurodegenerative movement disorder, and considerable progress has been made in understanding and treating the "typical" movement abnormalities of resting tremor, bradykinesia and rigidity. These cardinal PD features are all initially responsive to dopamine replacement therapy, and have been investigated intensively with respect to their relationships to degeneration of the nigrostriatal dopamine projection. More recently, increased attention has focused on the "non-motor" clinical aspects of PD, including cognitive, mood, chronobiological and peripheral autonomic defects. These clinical features are less reliably affected by dopaminergic therapy, and are likely to be associated with other, non-dopaminergic neural degenerations. Indeed, detailed postmortem assessments of PD brain reveal substantial neuronal losses in a variety of chemically-defined neurons, including brainstem serotonin and norepinephrine neurons and basal forebrain cholinergic neurons. Projects in the proposal will focus on dementia, depression, sleep-apnea and dysautonomia in PD patients, employing PET measures of presynaptic dopaminergic, serotoninergic and cholinergic CNS neurons and of peripheral sympathetic neurons. Results of the investigations may identify associations of non-motor PD signs and symptoms with the non-dopaminergic neuronal losses. These findings will establish additional therapeutic targets for symptomatic, but also for potential neuroprotective PD therapies. In addition, a majority of patients will be characterized with all 3 CNS PET measures. The availability of multiple markers of distinct neuronal populations involved in PD neurodegeneration will permit exploratory analyses to assess whether the degenerations are correlated (possibly manifestations of a common pathophysiology) or apparently independent (possibly a manifestation of multiple PD subtypes or pathophysiologies). Ultimately, better understanding of these non-motor features will be essential to developing future treatments that address the entire PD patient.

DETAILED DESCRIPTION:
Participating subjects may be eligible for one or more of the sub-projects that may have a focus on cognition, mood, sleep or autonomic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age 50 and above (40 for Normal Control population)
* diagnosed with PD
* Hoehn & Yahr 1-4,

Exclusion Criteria:

* other disorders which may resemble PD
* unstable medical conditions
* significant neurological or psychiatric disorders
* taking certain medications such as acetylcholinesterase inhibitors, neuroleptics, psychostimulants, tricyclic antidepressants,
* contraindication to MRI (pacemakers, metal in eye, etc)
* recent exposure to significant amount of ionizing radiation
* pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Movement Disorders Clinic, Hospital, Primary Care, Community
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To asses the non-motor aspects of PD | at initial visit and at 2 years for memory (PIB) and autonomic system symptoms (DTBZ and HED)
  The non-motor aspects that were studied included, sleep disorders, depression, memory, and autonomic system symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, M.D., Ph.D., Study Director — University of Michigan; Kirk Frey, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Zhou Z, Muller MLTM, Kanel P, Chua J, Kotagal V, Kaufer DI, Albin RL, Frey KA, Bohnen NI. Apathy rating scores and beta-amyloidopathy in patients with Parkinson disease at risk for cognitive decline. Neurology. 2020 Jan 28;94(4):e376-e383. doi: 10.1212/WNL.0000000000008683. Epub 2019 Nov 15. PMID 31732566